CLINICAL TRIAL: NCT01367327
Title: Effects of Therapeutic Music Combined With Loaded Sit-to-Stand Resistance Exercise for Children With Spastic Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0971762466; 98-2314-B-002-011-MY3 (Other Grant/Funding Number: NSC of ROC)
Record Dates: First submitted 2010-08-09; First posted 2011-06-07 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-02

CONDITIONS: Cerebral Palsy; Paraparesis, Spastic
Keywords: Exercise
MeSH Terms: conditions — Cerebral Palsy; Paraparesis, Spastic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise with music (Experimental): Loaded sit-to-stand exercise with music for 6 weeks
  Interventions: Behavioral: Loaded sit-to-stand exercise; Behavioral: Synchronized music
- Exercise without music (Active Comparator): Loaded sit-to-stand exercise without music for 6 weeks
  Interventions: Behavioral: Loaded sit-to-stand exercise

INTERVENTIONS:
Behavioral: Loaded sit-to-stand exercise — Loaded sit-to-stand exercise at home, 3 times a week for 6 weeks
Behavioral: Synchronized music — Synchronized music for loaded sit-to-stand exercise to guide movement
  Arms: Exercise with music

SUMMARY:
The purpose of study is to investigate the effects of PSE Music with a "home-based" loaded STS exercise program on the functional strength, gross motor function, daily participation, exercise involvement, motor control, and gait speed for children with spastic diplegia.

ELIGIBILITY:
Inclusion Criteria:

* children with SD, aged 5 to 13 year-old, and GMFCS level between I to III
* able to stand up from a chair independently and maintain standing for more than 2 seconds without falling
* able to follow verbal instructions

Exclusion Criteria:

* have orthopedic surgery, selective dorsal rhizotomy, or use of a baclofen pump within 6 months
* have orthopedic problems or other medical conditions preventing the child from joining the resistance exercise program, such as obvious LE joint contractures, uncontrolled epilepsy, or cardiopulmonary problems
* hearing loss or using hearing aid
* have mental disorders, such as pervasive developmental disorders and attention-deficit and disruptive behavior disorders

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure | 12 weeks

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory-Chinese Version | 12 weeks
Exercise Adherence and Volume | 12 weeks
Motor Control Variables of the STS Movement | 12 weeks
Pediatric Evaluation of Disability Inventory | 12 weeks
One-repetition maximum of loaded sit-to-stand test | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hua-Fang Liao, MS, Study Chair — Institute of Physical Therapy, National Taiwan University
Locations (1):
- Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Background] Liao HF, Liu YC, Liu WY, Lin YT. Effectiveness of loaded sit-to-stand resistance exercise for children with mild spastic diplegia: a randomized clinical trial. Arch Phys Med Rehabil. 2007 Jan;88(1):25-31. doi: 10.1016/j.apmr.2006.10.006. PMID 17207671
- [Background] Peng YC, Lu TW, Wang TH, Chen YL, Liao HF, Lin KH, Tang PF. Immediate effects of therapeutic music on loaded sit-to-stand movement in children with spastic diplegia. Gait Posture. 2011 Feb;33(2):274-8. doi: 10.1016/j.gaitpost.2010.11.020. Epub 2010 Dec 24. PMID 21185725